CLINICAL TRIAL: NCT06153459
Title: CORD-CHD: Clamp OR Delay Among Neonates With Congenital Heart Disease
Brief Title: Cord Clamping Among Neonates With Congenital Heart Disease
Acronym: CORD-CHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carl Backes, MD (Other)
Collaborators: The George Washington University Biostatistics Center (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Emory University (Other); Boston Children's Hospital (Other); University of Bristol (Other); Geisinger Commonwealth School of Medicine (Unknown); Duke University (Other); Children's Hospital of Philadelphia (Other); Sharp Mary Birch Hospital for Women & Newborns (Other); Université de Montréal (Other)
Responsible Party: Sponsor-Investigator, Carl Backes, MD, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00003337; UG3HL166794 (NIH); UG3HL166799 (Other Grant/Funding Number: NHLBI)
Record Dates: First submitted 2023-11-12; First posted 2023-12-01 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Congenital Heart Disease (CHD)
Keywords: cord clamping; echocardiography (ECHO); congenital heart disease (CHD); CORD-CHD
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Delayed Cord Clamping at 30 Seconds (DCC-30) (Active Comparator): The umbilical cord will be clamped between 1 - <60 seconds following delivery, with a goal of around 30 seconds.
  Interventions: Procedure: Umbilical Cord Clamping at ~30 seconds
- Delayed Cord Clamping at 120 Seconds (DCC-120) (Active Comparator): The umbilical cord will be clamped at 60 - 180- seconds following delivery, with a goal of around 120 seconds.
  In the DCC-120 group, if there is concern for pregnant individual or baby and their doctor is not able to wait until at least 60 seconds, the doctor may do cord milking, which is four gentle squeezes of the umbilical cord pushing blood from the placenta to baby.
  Interventions: Procedure: Umbilical Cord Clamping at ~120 seconds; Procedure: Umbilical Cord Milking

INTERVENTIONS:
Procedure: Umbilical Cord Clamping at ~30 seconds — Care team will wait to clamp the umbilical between 1-<60 seconds after birth. 30 seconds is the ideal time of clamping.
  Other Names: Randomized to DCC-30 Group
  Arms: Delayed Cord Clamping at 30 Seconds (DCC-30)
Procedure: Umbilical Cord Clamping at ~120 seconds — Care team will wait to clamp the umbilical cord between 60-180 seconds after birth.120 seconds is the ideal time of clamping
  Other Names: Randomized to DCC-120 Group
  Arms: Delayed Cord Clamping at 120 Seconds (DCC-120)
Procedure: Umbilical Cord Milking — For infants who need their cord clamped before the target in the DCC-120 group. Care team may milk the umbilical cord towards the infant four times. Cord milking should NOT be performed if the delay meets or exceeds 60 seconds.
  Umbilical cord milking will not be provided among participant-infant dyads in the DCC-30 group.
  Arms: Delayed Cord Clamping at 120 Seconds (DCC-120)

SUMMARY:
The goal of this clinical trial is to compare 2 different timepoints for clamping the umbilical cord at birth for term-born infants with a prenatal diagnosis of congenital heart disease (CHD). The main questions it aims to answer are:

* Does Delayed Cord Clamping at 120 seconds (DCC-120) or Delayed Cord Clamping at 30 seconds (DCC-30) after birth lead to better health outcomes?
* Does DCC-120 seconds or DCC-30 seconds after birth lead to better neuromotor outcomes at 22-26 months of infant age (postnatal)?

Participants will be asked to do the following:

* Participate in either DCC-120 or DCC-30 at birth (randomized assignment).
* Complete General Movements Assessment (GMA) at 3-4 months of infant age (postnatal), complete questionnaires / surveys at this time.
* Complete questionnaires / surveys at 9-12 months of infant age (postnatal).
* Complete Hammersmith Infant Neurological Examination (HINE), Developmental Assessment of Young Children 2 Edition (DAYC-2), and questionnaires / surveys at 22-26 months of infant age (postnatal).
* Permit data collection from electronic medical records for both the mother and infant study participants.

Investigators will compare DCC-120 vs. DCC-30 to see which approach is more beneficial to both the mother and baby with CHD.

DETAILED DESCRIPTION:
* AIM 1: Test the hypothesis that, among neonates with prenatally diagnosed significant CHD (ranking of 3 - 6 on the Fetal Cardiovascular Disease Severity Score [FCDSS]), DCC-120 results in lower global rank score (GRS), indicative of better health outcomes, compared with DCC-30.
* AIM 2: Test the hypothesis that, among neonates with prenatally diagnosed significant CHD (ranking from 3 - 6 on the Fetal Cardiovascular Disease Severity Score [FCDSS]), DCC-120 will result in better neuromotor outcomes at 22-26 months postnatal than DCC-30.

ELIGIBILITY:
Inclusion criteria are listed below and will be confirmed prior to randomization:

1. Fetal diagnosis of congenital heart disease (CHD) by prenatal ultrasound / echocardiography from local fetal ECHO, conducted on or after 18 weeks of gestation and prior to randomization. The study fetal diagnosis of CHD must be rated as 3 - 6 on the Fetal Cardiovascular Disease Severity Score (FCDSS), as determined by independent evaluators at the CORD-CHD trial ECHO Core at the Children's Hospital of Philadelphia (to determine final FCDSS eligibility for randomization).

   For each potential participant that has provided consent, the most relevant diagnostic prenatal ultrasound will be uploaded (shared) between 32 weeks of gestation and randomization for review by the ECHO Core. The ECHO Core will make the final FCDSS determination for eligibility status and stratification assignment.]

   [NOTE: A fetal diagnosis of CHD rated as 3 - 6 FCDSS per local review, including borderline cases, will be used to determine preliminary eligibility for consent. Among borderline cases, eligible patients will be included if there is a reasonable expectation of the need for surgery or cardiac catheterization during the birth hospitalization.]
2. Singleton gestation.
3. Gestational age at randomization for impending deliveries between 37 0/7 - 41 6/7 weeks of gestation inclusive based on clinical information and evaluation of the earliest ultrasound determined using criteria proposed by the American Congress of Obstetricians and Gynecologists (ACOG), the American Institute of Ultrasound in Medicine and the Society for Maternal-Fetal Medicine.

   [NOTE: Pregnant individuals who were admitted to the delivery hospital prior to 37 0/7 weeks of gestation remain eligible to randomize, provided they deliver within the 37 0/7 and 41 6/7 weeks "eligibility window". Alternatively, if an eligible dyad is randomized at or just prior to 41 6/7 weeks, they remain in trial.]
4. Consent for the participant and their infant

Exclusion criteria are listed below and will be confirmed prior to randomization:

Exclusion Criteria for Pregnant Individuals:

1. Pregnant individual is a gestational carrier or surrogate.
2. Compromise of the pregnant individual (e.g., vasa previa, placental accreta with hypotension, placental abruption, amniotic fluid embolism, uterine rupture, uterine inversion, disseminated intravascular coagulation), as determined by local care team

[NOTE: There is no limitation on pregnant individual's age]

Fetal Exclusion Criteria:

1. Fetal demise or planned termination of pregnancy prior to randomization
2. Tachyarrhythmia requiring transplacental therapy
3. Fetal hydrops, severe
4. Planned fetal surgery
5. Diaphragmatic hernia, omphalocele, gastroschisis, intestinal atresia
6. Major chromosomal defects (e.g., Trisomy 13, 18) identified prenatally; Trisomy 21 is allowed
7. Disease or disorder impacting candidacy for neonatal cardiac interventions
8. Parents choosing to limit treatment

Pregnancy Exclusion Criteria:

1. Delivery planned at an institution not affiliated with or does not refer to a CORD-CHD participating site
2. Participation in another prenatal interventional study that influences cord clamping or perinatal morbidity or mortality

Ages: 37 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Global Rank Score (Infant participant) | Up to 30 days post-discharge following congenital heart disease intervention
  Mortality=97;Heart transplant=96;Complication preventing cardiac intervention=95;Pre or Post-intervention neurologic complication=95;Pre or Post-intervention respiratory failure w/tracheostomy=95;Renal failure permanent dialysis=95;Unplanned cardiac surgery after initial cardiac intervention=94;Cardiac arrest=94;Pre or Post-intervention multisystem organ failure=94;Mechanical circulatory support=94;Pre-intervention polycythemia w/exchange transfusion/hemodilution=93;Unplanned cardiac catheterization after initial cardiac intervention=93;Pre-intervention mechanical ventilation=93;Pre-intervention necrotizing enterocolitis(Bell's II/III)=93;Pre-intervention shock=93;Pre-intervention unplanned hospitalization=93;Post-intervention bleeding reoperation=93;Delayed sternal closure=93;Pre-intervention renal failure temporary dialysis=93;Post-intervention renal failure, temporary dialysis=92;Post-intervention mechanical ventilation >7 days=92;Hospital length of stay >90 days=91,1-90 days=1-90

SECONDARY OUTCOMES:
Neuromotor Outcomes at 3-4 months of age (Infant participant) | 3-4 months after birth
  General Movements Assessment (GMA): The General Movements Assessment is used to identify absent or abnormal general movements in infants. General movements are spontaneous movements exhibited during fetal development and through the first 6 months of life after birth. Trained investigators will evaluate the infants general movements as: 1) Fidgety present; 2) Fidgety abnormal; and 3) Absent fidgety where "Fidgety present" is considered normal, and the other two outcomes are considered abnormal.
Impact of infant's congenital heart disease (Parents / Caregivers) | 3-4 months after birth
  Questionnaire/Survey on the impact of infant's congenital heart disease upon the family dynamic; Impact on Family Scale - Revised: The Impact on Family Scale - Revised is a questionnaire for parents / caregivers used to evaluate perceptions of the impact of an infant's chronic medical condition (e.g., congenital heart disease) upon the family. The IFS-R uses a 4-point Likert-type scale (strongly agree to strongly disagree) for responses. High scores correlate with parental / caregiver stressors and psychiatric symptoms, poor infant health, and increased pediatric hospitalizations and/or health maintenance requirement, representing worse outcomes.
Impact of infant's congenital heart disease (Parents / Caregivers) | 3-4 months after birth
  Questionnaire/Survey on the impact of infant's congenital heart disease upon the family dynamic; Functional Status II - Revised, Short Form: The Functional Status II - Revised, Short Form will be used to evaluate the functional status of infants that have been diagnosed with and undergone treatment for congenital heart disease. This survey, completed by parents / caregivers, is used to evaluate a core of 14 items using a 3-point Likert scale. The respondent (parent / caregiver) first rates the extent of difficulty with specific behaviors that the infant experiences, and then rates for those behaviors with difficulty, the extent to which the difficulty is due to the infants chronic illness. Higher scores generally indicate a reduced burden of chronic heart disease impacting the family, and therefore, a better outcome.
Impact of infant's congenital heart disease (Parents / Caregivers) | 9-12 months after birth
  Questionnaire/Survey on the impact of infant's congenital heart disease upon the family dynamic; Impact on Family Scale - Revised: The Impact on Family Scale - Revised is a questionnaire for parents / caregivers used to evaluate perceptions of the impact of an infant's chronic medical condition (e.g., congenital heart disease) upon the family. The IFS-R uses a 4-point Likert-type scale (strongly agree to strongly disagree) for responses. High scores correlate with parental / caregiver stressors and psychiatric symptoms, poor infant health, and increased pediatric hospitalizations and/or health maintenance requirement, representing worse outcomes.
Impact of infant's congenital heart disease (Parents / Caregivers) | 9-12 months after birth
  Questionnaire/Survey on the impact of infant's congenital heart disease upon the family dynamic; Functional Status II - Revised, Short Form: The Functional Status II - Revised, Short Form will be used to evaluate the functional status of infants that have been diagnosed with and undergone treatment for congenital heart disease. This survey, completed by parents / caregivers, is used to evaluate a core of 14 items using a 3-point Likert scale. The respondent (parent) first rates the extent of difficulty with specific behaviors that the infant experiences, and then rates for those behaviors with difficulty, the extent to which the difficulty is due to the infants chronic illness. Higher scores generally indicate a reduced burden of chronic heart disease impacting the family, and therefore, a better outcome.
Impact of infant's congenital heart disease (Parents / Caregivers) | 22-26 months after birth
  Questionnaire/Survey on the impact of infant's congenital heart disease upon the family dynamic; Impact on Family Scale - Revised: The Impact on Family Scale - Revised is a questionnaire for parents / caregivers used to evaluate perceptions of the impact of an infant's chronic medical condition (e.g., congenital heart disease) upon the family. The IFS-R uses a 4-point Likert-type scale (strongly agree to strongly disagree) for responses. High scores correlate with parental / caregiver stressors and psychiatric symptoms, poor infant health, and increased pediatric hospitalizations and/or health maintenance requirement, representing worse outcomes.
Impact of infant's congenital heart disease (Parents / Caregivers) | 22-26 months after birth
  Questionnaire/Survey on the impact of infant's congenital heart disease upon the family dynamic; Functional Status II - Revised, Short Form: The Functional Status II - Revised, Short Form will be used to evaluate the functional status of infants that have been diagnosed with and undergone treatment for congenital heart disease. This survey, completed by parents / caregivers, is used to evaluate a core of 14 items using a 3-point Likert scale. The respondent (parent) first rates the extent of difficulty with specific behaviors that the infant experiences, and then rates for those behaviors with difficulty, the extent to which the difficulty is due to the infants chronic illness. Higher scores generally indicate a reduced burden of chronic heart disease impacting the family, and therefore, a better outcome.
Neurodevelopmental Outcomes at 22-26 months (Infant participant) | 22-26 months after birth
  Hammersmith Infant Neurological Exam (HINE): The Hammersmith Infant Neurological Examination (HINE) consists of 26 items that assess different aspects of infant neurological function. The maximal global (total) score is 78, divided among the following domains: cranial nerve function (maximum score 15); posture (maximum score 18); movements (maximum score 6); muscle tone (maximum score 24) and reflexes and reactions (maximum score 15). Higher scores indicate better expected outcomes.
Neurodevelopmental Outcomes at 22-26 months (Infant participant) | 22-26 months after birth
  Developmental Assessment of Young Children, 2nd Edition (DAYC-2): The Developmental Assessment of Young Children, Second Edition (DAYC-2) is used to evaluate infants and children over 5 domains: cognition; communication; social-emotional development; physical development; and adaptive behavior. The DAYC-2 uses a norm-referenced sample to establish standardized scores in each domain, allowing investigators to compare the results to infants of similar age. Percentile ranks, and age equivalents are provided for each domain. Elements are graded on a simple "Yes" or "No" scale, with "Yes" being 1 point and "No" being 0 points. In general, higher scores reflect better expected outcomes.
Parental perspectives of outcomes (Parents / Caregivers) | 22-26 months after birth
  Survey of parent / caregiver opinions of expectations and outcomes as it relates to their infant with congenital heart disease. This questionnaire will examine parental perspectives with regards to health and neurodevelopmental outcomes, as compared to those commonly used in pediatric medicine. For example, parents / caregivers may place greater emphasis upon their child being able to conduct physical activity as compared to how well they perform tasks (fine and gross neuromotor function). Additionally, parents may express concern for their infant being able to eat without requiring a feeding tube, or breathing without the need for assistance or additional oxygen support. The survey will also seek to determine areas in which parents / caregivers feel there is room for improvement as it applies to their infant. There is no formal "scale" for this survey, as responses are primarily open-ended, requiring descriptive content analysis.
Delivery Complications and Outcomes (Pregnant individual participant) | Through hospital discharge (up to 1 month)
  Incidence of postpartum hemorrhage (defined as blood loss >1L within 24 hours post-delivery)
Delivery Complications and Outcomes (Pregnant individual participant) | Through hospital discharge (up to 1 month)
  Incidence of prolonged 3rd stage of labor (defined as retention of placenta for >30 minutes postpartum)
Delivery Complications and Outcomes (Pregnant individual participant) | Through hospital discharge (up to 1 month)
  Incidence of use of medications for postpartum hemorrhage management other than oxytocin (e.g., methergine, tranexamic acid, hemabate, misoprostol)
Delivery Complications and Outcomes (Pregnant individual participant) | Through hospital discharge (up to 1 month)
  Incidence of requirement for uterine balloon tamponade or other surgical intervention to treat postpartum hemorrhage
Delivery Complications and Outcomes (Pregnant individual participant) | Through hospital discharge (up to 1 month)
  Incidence of requirements for manual placental removal
Delivery Complications and Outcomes (Pregnant individual participant) | Through hospital discharge (up to 1 month)
  Incidence of requirement for transfusion, post-partum
Delivery Complications and Outcomes (Pregnant individual participant) | Through hospital discharge (up to 1 month)
  Volume of transfusion required, if applicable
Delivery Complications and Outcomes (Pregnant individual participant) | Through hospital discharge (up to 1 month)
  Type of transfusion required (e.g., whole blood, red blood cells, platelets, etc.), if applicable
Delivery Complications and Outcomes (Pregnant individual participant) | Through hospital discharge (up to 1 month)
  Incidence of postpartum endometritis
Delivery Complications and Outcomes (Pregnant individual participant) | Through hospital discharge (up to 1 month)
  Incidence of mortality

CONTACTS AND LOCATIONS:
Overall Officials: Carl Backes, MD, Principal Investigator — Nationwide Children's Hospital; Anup Katheria, MD, Principal Investigator — Sharp Mary Birch Hospital for Women & Newborns; Kevin Hill, MD, Principal Investigator — Duke Children's Hospital; Madeline Rice, PhD, Principal Investigator — George Washington University Biostatistics Center; Grecio (Greg) Sandoval, PhD, Principal Investigator — George Washington University Biostatistics Center; Scott Evans, PhD, Principal Investigator — George Washington University Biostatistics Center
Locations (21):
- United States (18):
  - Children's of Alabama, Birmingham, Alabama
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford, Palo Alto, California
  - Sharp Mary Birch Hospital for Woman and Newborns, San Diego, California
  - UF Health Shands Children's Hospital, Gainesville, Florida
  - Johns Hopkins Children's Center, Baltimore, Maryland
  - Children's of Mississippi, Jackson, Mississippi
  - The Children's Mercy Hospital, Kansas City, Missouri
  - SSM Health Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Duke Children's Hospital & Health Center, Durham, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Columbia, South Carolina
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
- Canada (3):
  - Stollery Children's Hospital, University of Alberta, Edmonton, Alberta
  - IWK Health Centre, Halifax, Nova Scotia
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available per NIH/NHLBI requirements (National Heart, Lung, and Blood Institute)
Supporting Information: SAP
Time Frame: 2 years after primary publication
Access Criteria: An archived dataset with documentation will be made available for additional uses by outside investigators, in collaboration with the study investigators. We will work with NIH/NHLBI program staff to develop a broad data sharing plan over time.

REFERENCES:
- [Background] Marzec L, Zettler E, Cua CL, Rivera BK, Pasquali S, Katheria A, Backes CH. Timing of umbilical cord clamping among infants with congenital heart disease. Prog Pediatr Cardiol. 2020 Dec;59:101318. doi: 10.1016/j.ppedcard.2020.101318. Epub 2020 Oct 28. PMID 34113067
- [Background] Backes CH, Huang H, Cua CL, Garg V, Smith CV, Yin H, Galantowicz M, Bauer JA, Hoffman TM. Early versus delayed umbilical cord clamping in infants with congenital heart disease: a pilot, randomized, controlled trial. J Perinatol. 2015 Oct;35(10):826-31. doi: 10.1038/jp.2015.89. Epub 2015 Jul 30. PMID 26226244
- [Background] Fite EL, Rivera BK, McNabb R, Smith CV, Hill KD, Katheria A, Maitre N, Backes CH. Umbilical cord clamping among infants with a prenatal diagnosis of congenital heart disease. Semin Perinatol. 2023 Jun;47(4):151747. doi: 10.1016/j.semperi.2023.151747. Epub 2023 Mar 18. No abstract available. PMID 37002126